CLINICAL TRIAL: NCT02614131
Title: Single-Dose and Multiple-Dose, Dose-Escalation Study With LY2599666 to Evaluate the Safety, Pharmacokinetics, and Tolerability in Healthy Subjects and Patients With Mild Cognitive Impairment Due to Alzheimer's Disease and Mild-to-Moderate Alzheimer's Disease
Brief Title: A Study of LY2599666 in Healthy Participants and Participants With Mild Cognitive Impairment or Alzheimer's Disease (AD)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: New data suggests that insufficient target engagement would be achieved for efficacy.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15491; I2L-MC-ALCA (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-11-23; First posted 2015-11-25 (Estimated); Results first posted 2019-09-23 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Healthy; Alzheimer's Disease; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — solanezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- LY2599666 (Part A) (Experimental): LY2599666 given subcutaneously (SC) once.
  Interventions: Drug: LY2599666
- Placebo (Part A) (Placebo Comparator): Placebo matching LY2599666 given SC once.
  Interventions: Drug: Placebo SC
- LY2599666 (Part B) (Experimental): LY2599666 given SC once weekly for 12 weeks (13 doses).
  Interventions: Drug: LY2599666
- Placebo (Part B) (Placebo Comparator): Placebo given SC once weekly for 12 weeks (13 doses).
  Interventions: Drug: Placebo SC
- Solanezumab (Part C) (Experimental): Solanezumab given intravenously (IV) once weekly or once every 4 weeks for 12 weeks.
  Interventions: Drug: Solanezumab
- Placebo (Part C) (Placebo Comparator): Placebo given IV once weekly or once every 4 weeks for 12 weeks.
  Interventions: Drug: Placebo IV

INTERVENTIONS:
Drug: LY2599666 — Administered SC
  Arms: LY2599666 (Part A); LY2599666 (Part B)
Drug: Solanezumab — Administered IV
  Other Names: LY2062430
  Arms: Solanezumab (Part C)
Drug: Placebo SC — Administered SC
  Arms: Placebo (Part A); Placebo (Part B)
Drug: Placebo IV — Administered IV
  Arms: Placebo (Part C)

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of the study drug known as LY2599666 in different groups of people - those who are healthy, those who have mild cognitive impairment due to Alzheimer's Disease (AD), and those with mild-to-moderate AD. The study will measure how much LY2599666 gets into the bloodstream and how long it takes the body to get rid of it. It will also evaluate how LY2599666 affects the body. The study has three parts. Part A will last about 2 months. Parts B and C will each last about 23 weeks. Participants may only enroll in one part.

ELIGIBILITY:
Inclusion Criteria:

Healthy Participants Part A:

* Overtly healthy males or females as determined by medical history and physical examination
* Have a body mass index (BMI) between 18.0 and 32.0 kilograms per meter squared (kg/m²), inclusive

Participants With Mild Cognitive Impairment or Alzheimer's Disease (AD) [Part B and C]:

* Participants are at least 50 years old at screening
* Present with Mild Cognitive Impairment (MCI) due to Alzheimer's Disease (AD) or mild-to-moderate AD
* Have a caregiver/study informant who provides a separate written informed consent to participate
* Have adequate vision and hearing for neuropsychological testing in the opinion of the investigator
* Positive florbetapir scan

Exclusion Criteria:

All Participants

* Are currently enrolled in a clinical trial involving an investigational product or off-label use of a drug or device or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have known allergies to LY2599666, solanezumab, or any related compounds or components of the formulations, or have a history of significant atopy
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study
* Have an abnormal blood pressure as determined by the investigator
* Have significant allergies to humanized monoclonal antibodies, diphenhydramine, epinephrine, or methylprednisone
* Require treatment with other monoclonal antibodies

Participants With Mild Cognitive Impairment or Alzheimer's Disease (AD) [Part B and C]

* Have medical or surgical conditions in which lumbar puncture and or/catheter insertion is contraindicated
* Have any contraindication for magnetic resonance imaging (MRI) studies, including claustrophobia, the presence of metal (ferromagnetic) implants, or a cardiac pacemaker that is not compatible with MRI

Participants With Mild Cognitive Impairment or Alzheimer's Disease (AD) [Part C]

* Have had lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years, cervical carcinoma in situ, or in situ prostate cancer with a normal prostate-specific antigen post treatment

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- United States (3):
  - Parexel Early Phase Unit at Glendale, Glendale, California
  - CRI Lifetree, Marlton, New Jersey
  - PRA Health Sciences, Salt Lake City, Utah
- Japan (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Kobe
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Shinjuku-Ku

REFERENCES:
- See also: A Study of LY2599666 in Participants With Mild Cognitive Impairment or Alzheimer's Disease (AD) — https://trials.lillytrialguide.com/en-US/trial/3BploURamQkS2qACASCoSc#?postal=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Following the enrollment of 7 participants into Part B Cohort 5, a decision was made to stop the development of LY2599666 based on the lack of efficacy results of another compound directed against the same target. Participants were not enrolled for Part B Cohorts 6 and 7 or Part C Cohorts 8 and 9.
Groups:
- Placebo (Part A - Healthy Participants): Placebo matching dose given subcutaneously (SC) once.
- 10 mg LY2599666 (Part A Cohort 1): 10 mg LY2599666 given SC once.
- 25 mg LY2599666 (Part A Cohort 2): 25 mg LY2599666 given SC once.
- 100 mg LY2599666 (Part A Cohort 3): 100 mg LY2599666 given SC once.
- 200 mg LY2599666 (Part A Cohort 4): 200 mg LY2599666 given SC once.
- Placebo (Part B - Cognitively Impaired): Placebo matching dose given SC.
- 25 mg LY2599666 (Part B Cohort 5): 25 mg LY2599666 given SC once weekly for 12 weeks (13 doses).
Period: Overall Study
Arm/Group | Placebo (Part A - Healthy Participants) | 10 mg LY2599666 (Part A Cohort 1) | 25 mg LY2599666 (Part A Cohort 2) | 100 mg LY2599666 (Part A Cohort 3) | 200 mg LY2599666 (Part A Cohort 4) | Placebo (Part B - Cognitively Impaired) | 25 mg LY2599666 (Part B Cohort 5)
Started | 11 | 8 | 8 | 8 | 8 | 2 | 5
Received at Least One Dose of Drug | 11 | 8 | 8 | 8 | 8 | 2 | 5
Completed | 10 | 8 | 8 | 8 | 8 | 2 | 4
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Placebo (Part A): Placebo matching dose given subcutaneously (SC) once.
- Placebo (Part B): Placebo matching dose given SC.
- Total: Total of all reporting groups
Arm/Group | Placebo (Part A) | 10 mg LY2599666 (Part A Cohort 1) | 25 mg LY2599666 (Part A Cohort 2) | 100 mg LY2599666 (Part A Cohort 3) | 200 mg LY2599666 (Part A Cohort 4) | Placebo (Part B) | 25 mg LY2599666 (Part B Cohort 5) | Total
Number analyzed (Participants) | 11 | 8 | 8 | 8 | 8 | 2 | 5 | 50
Age, Customized [Mean (Standard Deviation); unit: years] — Population: All randomized participants in Part A and Part B.
  years
    Part A: number analyzed (Participants) | 11 | 8 | 8 | 8 | 8 | 0 | 0 | 43
    Part A | 45.8 (10.7) | 40.0 (14.1) | 41.1 (13.5) | 38.9 (12.9) | 44.4 (16.2) |  |  | 42.3 (13.0)
    Part B: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 2 | 5 | 7
    Part B |  |  |  |  |  | 67 (12.7) | 69 (5.3) | 68.4 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 1 | 1 | 3 | 1 | 3 | 14
  Male | 9 | 5 | 7 | 7 | 5 | 1 | 2 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 1 | 3 | 1 | 0 | 0 | 9
  Not Hispanic or Latino | 9 | 6 | 7 | 5 | 7 | 2 | 5 | 41
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 5 | 3 | 3 | 3 | 3 | 1 | 2 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 1 | 1 | 1 | 1 | 0 | 0 | 8
  White | 2 | 4 | 4 | 4 | 4 | 1 | 3 | 22
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 8 | 8 | 8 | 8 | 1 | 3 | 47
  Japan | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event (SAE) Considered by the Investigator to be Related to Study Drug Administration
Description: Number of participants who experienced one or more treatment-emergent serious adverse events related to study treatment. A summary of other non-serious AEs, and all SAE's, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline through 4 weeks (Part A) or 16 weeks (Part B )
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Part A) | 10 mg LY2599666 (Part A Cohort 1) | 25 mg LY2599666 (Part A Cohort 2) | 100 mg LY2599666 (Part A Cohort 3) | 200 mg LY2599666 (Part A Cohort 4) | Placebo (Part B) | 25 mg LY2599666 (Part B Cohort 5)
Number analyzed (Participants) | 11 | 8 | 8 | 8 | 8 | 2 | 5
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY2599666 Part A
Description: PK: Cmax of LY2599666 after a single dose administered subcutaneously.
Time Frame: Day 1: Pre-dose and 2, 4, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264, 336, 504, 672 hours post-dose (Part A)
Population: All participants who received at least one dose of study drug in Part A and had evaluable Cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | 10 mg LY2599666 (Part A Cohort 1) | 25 mg LY2599666 (Part A Cohort 2) | 100 mg LY2599666 (Part A Cohort 3) | 200 mg LY2599666 (Part A Cohort 4)
Number analyzed (Participants) | 8 | 8 | 8 | 8
nanograms per milliliter (ng/mL) | NA (NA) — Majority of samples for 10 mg LY2599666 arm were below the limit of quantification in concentration and Cmax summary was not able to be calculated. | 780 (74) | 5310 (28) | 9810 (44)

3. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY2599666 Part B
Description: PK: Cmax of LY2599666 after multiple doses administered subcutaneously.
Time Frame: Day 85: Pre-dose, 2, 4, 8, 12, 24, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 96, 120, 168, 216, 264, 336, 504, 672 hours post-dose (Part B)
Population: All participants who received at least one dose of drug in Part B and had evaluable Cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- 25 mg LY2599666 (Part B Cohort 5): 25 mg LY2599666 given SC once weekly.
Arm/Group | 25 mg LY2599666 (Part B Cohort 5)
Number analyzed (Participants) | 4
ng/mL | 636 (41)

4. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC 0-∞) of LY2599666 Part A
Description: Area Under the Concentration versus Time Curve of zero to infinity (0 to ∞) after a single dose of LY2599666 administered subcutaneously.
Time Frame: Day 1: Pre-dose and 2, 4, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264, 336, 504, 672 hours post-dose (Part A)
Population: All participants who received at least one dose of drug in Part A and had evaluable AUC data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter (ng*hr/mL)
Arm/Group | 10 mg LY2599666 (Part A Cohort 1) | 25 mg LY2599666 (Part A Cohort 2) | 100 mg LY2599666 (Part A Cohort 3) | 200 mg LY2599666 (Part A Cohort 4)
Number analyzed (Participants) | 8 | 8 | 8 | 8
nanograms*hour per milliliter (ng*hr/mL) | NA (NA) — Majority of samples for 10 mg LY2599666 arm were below the limit of quantification in concentration and AUC summary was not able to be calculated. | 96200 (30) | 691000 (20) | 1590000 (27)

5. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Zero to 168 Hours (AUC 0-168) of LY2599666 Part B
Description: Area Under the Concentration time versus curve from 0-168 hours after weekly dose of LY2599666 administered subcutaneously.
Time Frame: Day 85: Pre-dose, 2, 4, 8, 12, 24, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 96, 120, 168 hours post-dose (Part B)
Population: All participants who received at least one dose of drug in Part B and had evaluable AUC data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- 25 mg LY2599666 (Part B Cohort 5) Day 85: 25 mg LY2599666 given SC once weekly.
Arm/Group | 25 mg LY2599666 (Part B Cohort 5) Day 85
Number analyzed (Participants) | 4
ng*hr/mL | 76100 (30)

6. Secondary Outcome: Plasma Amyloid Beta1-40 (Aβ1-40 ) Concentration Part A
Description: Concentration of plasma amyloid beta 1-40 in healthy participants after single dose of LY2599666 administered subcutaneously.
Time Frame: Day 1: Pre-dose and 2, 4, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264, 336, 504, 672 hours post-dose (Part A)
Population: All participants who received at least one dose of study drug in Part A and had evaluable Aβ1-40 data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picograms per milliliter (pg/mL)
Arm/Group | 10 mg LY2599666 (Part A Cohort 1) | 25 mg LY2599666 (Part A Cohort 2) | 100 mg LY2599666 (Part A Cohort 3) | 200 mg LY2599666 (Part A Cohort 4)
Number analyzed (Participants) | 8 | 8 | 8 | 8
picograms per milliliter (pg/mL) | 18800 (29) | 36200 (13) | 49500 (10) | 67700 (20)

7. Secondary Outcome: Plasma Amyloid Beta (Aβ1-40 and Aβ1-42) Concentration Part B
Description: Concentration of plasma amyloid beta 1-40 and 1-42, in participants with Mild Cognitive Impairment (MCI) or Alzheimer Disease, after multiple doses of LY2599666 administered subcutaneously.
Time Frame: as for outcome 3
Population: All participants who received at least one dose of study drug in Part B and had evaluable Aβ1-40 or Aβ1-42 data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | 25 mg LY2599666 (Part B Cohort 5)
Number analyzed (Participants) | 4
pg/mL
  Aβ1-40 | 51400 (14)
  Aβ1-42 | 5730 (10)

ADVERSE EVENTS:
Time Frame: Part A up to 29 days and Part B up to 113 days
Description: All participants who received at least one dose of study drug.
Arm/Group | Placebo (Part A) | 10 mg LY2599666 (Part A Cohort 1) | 25 mg LY2599666 (Part A Cohort 2) | 100 mg LY2599666 (Part A Cohort 3) | 200 mg LY2599666 (Part A Cohort 4) | Placebo (Part B) | 25 mg LY2599666 (Part B Cohort 5)
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/8 | 0/8 | 0/8 | 0/8 | 0/2 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/8 | 0/8 | 0/8 | 0/8 | 0/2 | 1/5
Other Adverse Events (participants affected / at risk) | 2/11 | 4/8 | 3/8 | 2/8 | 5/8 | 2/2 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Part A) (N=11) | 10 mg LY2599666 (Part A Cohort 1) (N=8) | 25 mg LY2599666 (Part A Cohort 2) (N=8) | 100 mg LY2599666 (Part A Cohort 3) (N=8) | 200 mg LY2599666 (Part A Cohort 4) (N=8) | Placebo (Part B) (N=2) | 25 mg LY2599666 (Part B Cohort 5) (N=5)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Part A) (N=11) | 10 mg LY2599666 (Part A Cohort 1) (N=8) | 25 mg LY2599666 (Part A Cohort 2) (N=8) | 100 mg LY2599666 (Part A Cohort 3) (N=8) | 200 mg LY2599666 (Part A Cohort 4) (N=8) | Placebo (Part B) (N=2) | 25 mg LY2599666 (Part B Cohort 5) (N=5)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ocular discomfort (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faecal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (2)
Injection site haemorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vessel puncture site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (3)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Development of LY2599666 was stopped based on lack of efficacy of another compound directed against the same target. Following the enrollment of seven participants into Part B Cohort 5, enrollment was stopped.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days